CLINICAL TRIAL: NCT06178796
Title: Bone-Implant Contact Surface Influence on Dental Implant Stability in Fresh Extraction and Healed Sites
Brief Title: Bone-Implant Contact Surface Influence on Dental Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUDHF_CER_01
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Missing Teeth
Keywords: Dental implant, primary stability, immediate placement
MeSH Terms: conditions — Anodontia | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- With graft (Active Comparator)
  Interventions: Device: Dental implant
- Without graft (Active Comparator)
  Interventions: Device: Dental implant
- Delayed healing site (Active Comparator)
  Interventions: Device: Dental implant

INTERVENTIONS:
Device: Dental implant — Dental implant placement

SUMMARY:
This study aims to evaluate the changes in the stability and bone-implant contact surface of implants of the same macro-design placed with particle grafting in the fresh extraction socket, without grafting, and placed in healed implant sites.

ELIGIBILITY:
Inclusion Criteria:

* Having a non-repairable premolar or molar tooth, or an edentulous area where the corresponding teeth have been extracted at least six months ago,
* At least 18 years old,
* Maintaining good dental hygiene,
* Having a favorable occlusion,
* Having intact socket walls after extraction.

Exclusion Criteria:

* Any local or systemic disorders that had contraindications for dental implant insertion,
* Pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Implant Stability Quotient (ISQ) values | 12 weeks
  Implant Stability Quotient (ISQ) is a scale from 1 to 100, to quantify implant stability in bone (higher values mean higher stability). ISQ numerical values are generated by applying resonance frequency analysis (RFA) or sound waves through a specialized peg attached to the implant. Data were combined to reduce the number of intervals for analysis purposes. Data from intervals were combined as follows:
  T0: baseline T1: follow-up of eight weeks T2: follow-up of twelve weeks
Change in bone-implant contact surface | 12 weeks
  The tooth slated for extraction will be segmented from the preoperative CBCT data, followed by a virtual tooth extraction process. For each patient, intraoral surface scanning with the scanbodies in place will be conducted using an intraoral scanner. This datas will be overlaid onto the postoperative intraoral scan image. The area where the implant surface made contact with the extracted tooth surface will be identified as the surface without implant bone contact (BINC), while the remaining area will be designated the bone implant contact (BIC) surface. By subtracting the sum of the BINC and BIC from the entire implant surface, the implant surface facing the gap space (IGS) and its corresponding area on the BINC side will obtain. To isolate the BIC surface for measurement, the sum of the BINC and BIC from the sum of the BINC and IGS will subtracted. This result will then be added to the total implant surface measurement, divided by two, allowing for the measurement of the BIC surface.
Primary insertion torque value | 1 day At the implant placement
  The torque value was recorded as insertion torque value of this case at the moment when the implant positioned at the 1mm under the socket wall edge and correct hex position. It gives numerical values from 0 to 100 (higher values mean higher stability).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided